CLINICAL TRIAL: NCT01846039
Title: A Prospective, Open-label Study of the Safety and Efficacy of JUVÉDERM VOLUMA® to Enhance the Aesthetic Appearance of the Asian Nose
Brief Title: JUVÉDERM VOLUMA® to Enhance the Appearance of the Asian Nose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VOLXC-AP-ND-001
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Asian Nose Enhancement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JUVÉDERM VOLUMA® (Experimental): Participants treated with JUVÉDERM VOLUMA® up to 3 mLs administered by intradermal injection.
  Interventions: Device: Crosslinked hyaluronic acid gel

INTERVENTIONS:
Device: Crosslinked hyaluronic acid gel — Up to 3 mL administered by intradermal injection
  Other Names: JUVÉDERM VOLUMA®

SUMMARY:
A prospective, open-label, observational study of the safety and efficacy of JUVÉDERM VOLUMA® to enhance the aesthetic appearance of the Asian nose.

ELIGIBILITY:
Inclusion Criteria:

* Asian subjects aged 20 years of age or older with dissatisfaction of their aesthetic appearance due to structural features of their nose
* Subjects who, in the opinion of the Investigator, can achieve a clinically meaningful aesthetic correction of their nose with VOLUMA® treatment

Exclusion Criteria:

* -Subjects requiring filler treatment in or around the tip of the nose or between the eyebrows (glabellar region) to achieve a good aesthetic outcome
* prior nasal surgery, including grafts, implants or filler injection to the nose area
* Subjects with a history of sinusitis or rhinitis
* Subjects unlikely to achieve a meaningful aesthetic result with the prescribed dosage regimen of the study product.
* Subjects receiving botulinum toxin treatment for any indication within 3 months of the study or planning to receive botulinum toxin during the study
* Subjects who have previously received aesthetic treatment in the forehead, glabellar, and/or nose area with any dermal filler
* Subjects with a history of any significant adverse events caused by dermal fillers
* Subjects with a history of allergic responses to lidocaine or fillers
* Subjects who are pregnant or breastfeeding or wish to become pregnant during the study
* Subjects of child-bearing age who are not prepared to practice an adequate form of contraception during the course of the study
* Subjects with traumatic scars in the treatment area or a history of active inflammation, infection, cancerous lesion, or an unhealed wound in the treatment area
* Subjects requiring dental or oral surgery, including dental implants, during the study period
* Subjects with a history of bleeding disorders
* Subjects who are smokers
* Subjects using blood thinning products within 10 days of the screening visit
* Subjects with a history of connective tissue disease (e.g., rheumatoid arthritis, lupus, scleroderma, etc) causing skin scarring
* Subjects with a history of untreated epilepsy or other significant medical conditions
* Subjects with a history of alcoholism or drug abuse of dependence
* Subjects participating or likely to participate in another clinical trial within 30 days of screening or during the 1 year period of the study
* Subjects with any other medical condition, which in the opinion of the Investigator, might compromise the subject's ability to tolerate the injection procedure or comply with requirements of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2013-09-01 (Actual); Study Completion 2014-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Australia (2):
  - Sydney, New South Wales
  - Gold Coast, Queensland

REFERENCES:
- [Background] Liew S, Scamp T, de Maio M, Halstead M, Johnston N, Silberberg M, Rogers JD. Efficacy and Safety of a Hyaluronic Acid Filler to Correct Aesthetically Detracting or Deficient Features of the Asian Nose: A Prospective, Open-Label, Long-Term Study. Aesthet Surg J. 2016 Jul;36(7):760-72. doi: 10.1093/asj/sjw079. Epub 2016 Jun 14. PMID 27301371

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | JUVÉDERM VOLUMA®
Started | 29
Completed | 27
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Subject Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | JUVÉDERM VOLUMA®
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥ 1 Grade Improvement on the Assessment of Aesthetic Improvement Scale (AAIS) as Assessed by the Central Evaluating Physician at Day 113
Description: The independent central evaluating physician evaluated the improvement of the participant's nose as compared to Baseline using the AAIS 5-point scale: -2 (much worse) to +2 (much improved) at Day 113. The percentage of participants with a ≥ 1 grade improvement from Baseline is reported.
Time Frame: Baseline, Day 113
Population: Intent-to-treat population included all enrolled participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA®
Number analyzed (Participants) | 29
percentage of participants | 93.1

2. Primary Outcome: Percentage of Participants With a ≥ 1 Grade Improvement on the AAIS as Assessed by the Patient at Day 113
Description: The participant evaluated the improvement of their nose as compared to Baseline using the AAIS 5-point scale: -2 (much worse) to +2 (much improved) at Day 113. The percentage of participants with a ≥ 1 Grade Improvement from Baseline is reported.
Time Frame: Baseline, Day 113
Population: Intent-to-treat population included all enrolled participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA®
Number analyzed (Participants) | 29
percentage of participants | 93.1

3. Secondary Outcome: Percentage of Participants With a ≥ 1 Grade Improvement on the AAIS as Assessed by the Central Evaluating Physician
Description: The independent central evaluating physician evaluated the improvement of the participant's nose compared to Baseline using the AAIS 5-point scale: -2 (much worse) to +2 (much improved) at Days 239 and 421. The percentage of participants with a ≥ 1 grade improvement from Baseline is reported.
Time Frame: Baseline, Days 239 and 421
Population: Intent-to-treat population included all enrolled participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA®
Number analyzed (Participants) | 29
percentage of participants
  Day 239 | 100.0
  Day 421 | 96.6

4. Secondary Outcome: Percentage of Participants With a ≥ 1 Grade Improvement on the AAIS as Assessed by the Patient
Description: The participant evaluated the improvement of their nose as compared to Baseline using the AAIS 5-point scale: -2 (much worse) to +2 (much improved) at Days 239 and 421. The percentage of participants with a ≥ 1 grade improvement from Baseline is reported
Time Frame: Baseline, Days 239 and 421
Population: Intent-to-treat population included all enrolled participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA®
Number analyzed (Participants) | 29
percentage of participants
  Day 239 | 96.6
  Day 421 | 96.6

5. Secondary Outcome: Percentage of Participants Satisfied or Very Satisfied Based on the Nose Satisfaction Scale (NSS)
Description: Participants assessed their satisfaction with the appearance of their nose at Days 113, 239 and 421 using the NSS 5-point scale: -2 (very dissatisfied) to 2 (very satisfied). The percentage of participants who rated themselves as satisfied or very satisfied is reported.
Time Frame: Days 113, 239 and 421
Population: Intent-to-treat population included all enrolled participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA®
Number analyzed (Participants) | 29
percentage of participants
  Day 113 | 93.1
  Day 239 | 89.7
  Day 421 | 89.7

6. Secondary Outcome: Percentage of Participants Satisfied or Very Satisfied Based on the Treatment Satisfaction Scale (TSS)
Description: Participants assessed their satisfaction with the study drug (VOLUMA) treatment at Days 113, 239 and 421 using the TSS 5-point scale: -2 (very dissatisfied) to 2 (very satisfied). The percentage of participants satisfied or very satisfied with study drug treatment is reported.
Time Frame: Days 113, 239 and 421
Population: Intent-to-treat population included all enrolled participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA®
Number analyzed (Participants) | 29
percentage of participants
  Day 113 | 82.8
  Day 239 | 82.8
  Day 421 | 79.3

7. Secondary Outcome: Percentage of Participants Who Would Recommend VOLUMA Treatment of the Nose to Others
Time Frame: Days 113, 239 and 421
Population: Intent-to-treat population included all enrolled participants who received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA®
Number analyzed (Participants) | 29
percentage of participants
  Day 113 | 89.7
  Day 239 | 89.7
  Day 421 | 86.2

ADVERSE EVENTS:
Arm/Group | JUVÉDERM VOLUMA®
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 29/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JUVÉDERM VOLUMA® (N=29)
Injection site swelling (General disorders) | 28
Injection site erythema (General disorders) | 20
Injection site bruising (General disorders) | 16
Injection site pain (General disorders) | 11
Injection site discomfort (General disorders) | 8
Injection site hypoaesthesia (General disorders) | 2
Injection site reaction (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.